CLINICAL TRIAL: NCT02121730
Title: Identification of Key Risk Factors Associated With Neoplastic Complications After Renal Transplantation in Nord-Pas de Calais, Normandy and Picardy Regions
Brief Title: Identification of Risk Factors Associated With Neoplastic Complications After Renal Transplantation in Nord-Pas de Calais , Normandy and Picardy Regions
Acronym: FRISC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0006
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Cancer of Kidney
Keywords: grafting kidney; Cancer
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplantation: Patients who had undergone renal transplantation for 10 years in the interregion Northwest (Normandy, Picardy and Nord-Pas de Calais).

SUMMARY:
Kidney transplantation is now the treatment of choice for end-stage renal disease (ESRD). Between 2800 and 3000 kidney transplants are performed each year in France and more than 33 000 patients are living with a functioning graft.

Preventing allograft rejection requires the use of immunosuppressive therapy, the intensity decreases as the distance from the day of transplantation. Unfortunately, treatment favors certain complications, including infectious and neoplastic. These represent a major cause of mortality in these patients. If the frequency of skin cancer is greatly increased in this population, that of solid tumors remains a concern. Approximately 20% of patients develop cancer after 10 years of graft , half non- skin cancers, the main risk factor is immunosuppressive therapy .

The aim of the study is to evaluate, in a large population of patients treated in 4 regions ( the Nord-Pas de Calais, the Upper and Lower Normandy and Picardy) risk factors (in particular the nature of the immunosuppressive treatment) of developing a neoplastic complication, skin cancers and solid tumors, after renal transplantation.

DETAILED DESCRIPTION:
A retrospective analysis of the previous 10 years, from 2002 to 2011 will be conducted. This study will better understand the epidemiology of these complications but also allow to identify risk factors associated, including demographic, environmental and related to immunosuppressive therapy.

Thereafter, we hope to implement preventive measures or prospective studies, allowing us to reduce the prevalence of this complication.

ELIGIBILITY:
Inclusion Criteria:

* All adult renal transplant patients in the 4 centers of interregion North - West
* Patients transplanted during the period from 1 January 2002 and 31 December 2011
* Patients recipients of first, second or third renal transplantation
* Patients transplant recipients from a living or deceased donor whatever the immunological risk
* Eligible patients will be included after being informed by their doctor and after accepting their data to be processed in the framework of this study
* Patient with a health insurance coverage

Exclusion Criteria:

* Patients transplanted as child
* Patients transplanted before 1 January 2002
* Patients followed in the interregion but transplanted in another center
* Patients recipients of a double transplant (two kidneys or kidney plus other organ)
* Patients that do not accept their medical data to be included in the database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone renal transplantation for 10 years in the French interregion Northwest (Normandy, Picardy and Nord-Pas de Calais).
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2014-11-17 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Association between neoplastic complications and cancers | 10 years
  Correlation, in a population of renal transplant patients followed in interregion Northwest, of the association of neoplastic complications after renal transplantation, skin cancers and solid tumors outside the non-Hodgkin's lymphoma and the terms of immunosuppressive treatment used

SECONDARY OUTCOMES:
Risk factors | 10 years
  Identify the main risk factors for developing cancer after transplantation, besides immunosuppressive therapy
Incidence | 10 years
  Evaluate the incidence of neoplastic complications after renal transplantation in interregion Northwest
Typology of cancers | 10 years
  Assess the distribution and respective frequency of different types of cancer, skin and solid tumors in this group of patients
Survival prognosis | 10 years
  Establish the prognosis and survival of transplanted patients with a diagnosis of cancer after transplantation
Survival factors | 10 years
  Analyze the factors associated with the survival of transplanted patients who developed cancer after transplantation
Graft survival | 10 years
  Evaluate graft survival in the group of patients who develop post- transplantation cancer , especially after cancer diagnosis
Rejection number | 10 years
  Determine the number of cellular acute rejection and humoral rejections in patients who developed cancer and those free from this complication and analyze the prevalence of releases in the period following the diagnosis of cancer
Renal function after cancer | 10 years
  To analyze the evolution of renal function after cancer diagnosis
Cancer management | 10 years
  Analyze the management of these cancers, in particular as regards the strategy of immunosuppressive therapy after cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Choukroun, MD, PhD, Study Director — CHU Amiens; Marc Hazzan, MD, PhD, Study Chair — CHRU LILLE; Bruno Hurault de Ligny, MD, PhD, Study Chair — CHU CAEN; Michel Godin, MD, PhD, Study Chair — CHU Rouen
Locations (4):
- France (4):
  - CHU Amiens, Amiens
  - CHU CAEN, Caen
  - Chru Lille, Lille
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No